CLINICAL TRIAL: NCT03331666
Title: Impact of LDL-cholesterol Lowering on Platelet Activation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated Prematurely due to COVID-19
Sponsor: Columbia University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Nan Wang, Associate Professor of Medical Sciences (in Medicine) at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AAAR1041
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Familial Hypercholesterolemia
Keywords: Hyperlipidemia, Hypercholesterolemia, atherothrombosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipidemias; Hypercholesterolemia; Thrombosis | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evolocumab (Active Comparator): Subjects will start with placebo and will receive Evolocumab 140 mg every 14 days starting Day 14 until Day 196.
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): Subjects will start with placebo and will receive Evolocumab 140 mg every 14 days starting Day 28 until Day 196.
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — 140 mg every 14 days A monoclonal antibody designed for the treatment of hyperlipidemia
  Other Names: REPATHA

SUMMARY:
The primary goal is to assess the impact of Evolocumab therapy on platelet function of familial hypercholesterolemia (FH) patients in a randomized, double blind study. Evolocumab is a humanized monoclonal antibody that targets circulating PCSK9, increases hepatic LDL receptor, decreases plasma LDL cholesterol and reduces risk of cardiovascular events. Evolocumab (brand name Rapatha) has been approved by FDA along with diet and maximally tolerated statin therapy in adults with FH or atherosclerotic heart or blood vessel problems, who need additional lowering of LDL cholesterol.

The secondary goal is to determine if platelet activation or the response to Evolocumab therapy is modified by rs3184504 polymorphism. The investigators believe that these investigations will complement ongoing studies to demonstrate that Evolocumab reduces athero-thrombotic risk and aid the decision-making as to whether Evolocumab can reduce the atherothrombotic risk in acute coronary syndrome (ACS) patients.

DETAILED DESCRIPTION:
Hyperlipidemia as exemplified by familial hypercholesterolemia is associated with increased platelet activation and an underlying pro-coagulant state. Hyperlipidemia primes platelets and increases platelet activation in response to various agonists. Plasma cholesterol levels appear to have a critical role in modulating platelet activity as hypercholesterolemia increases platelet activation more potently than hypertriglyceridemia. Increased platelet reactivity may contribute to the increased risk of atherothrombosis associated with hypercholesterolemia. Plasma levels of platelet activation markers such as thrombin-antithrombin complex (TAT), soluble P-selectin (sP-selectin), soluble CD40L (sCD40L) or P-selectin exposure at surface of platelets are increased in hypercholesterolemic patients. Increased levels of the platelet activation markers are associated with increased platelet membrane cholesterol content in hypercholesterolemia.Statins may show antithrombotic properties.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a clinical diagnosis of familial hypercholesterolemia (FH)
* Subjects who are referred to Dr. Ginsberg's Lipid Practice for treatment with PCSK9 inhibitor
* Subjects with LDL cholesterol levels >100 mg/dl on baseline treatment with statins and/or ezetimibe

Exclusion Criteria:

* Children under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ginsberg, MD, Study Director — Columbia University; Nan Wang, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carvalho AC, Colman RW, Lees RS. Platelet function in hyperlipoproteinemia. N Engl J Med. 1974 Feb 21;290(8):434-8. doi: 10.1056/NEJM197402212900805. No abstract available. PMID 4359434
- [Background] CONNOR WE, HOAK JC, WARNER ED. Massive thrombosis produced by fatty acid infusion. J Clin Invest. 1963 Jun;42(6):860-6. doi: 10.1172/JCI104778. No abstract available. PMID 14022629
- [Background] Owens AP 3rd, Passam FH, Antoniak S, Marshall SM, McDaniel AL, Rudel L, Williams JC, Hubbard BK, Dutton JA, Wang J, Tobias PS, Curtiss LK, Daugherty A, Kirchhofer D, Luyendyk JP, Moriarty PM, Nagarajan S, Furie BC, Furie B, Johns DG, Temel RE, Mackman N. Monocyte tissue factor-dependent activation of coagulation in hypercholesterolemic mice and monkeys is inhibited by simvastatin. J Clin Invest. 2012 Feb;122(2):558-68. doi: 10.1172/JCI58969. Epub 2012 Jan 3. PMID 22214850
- [Background] Harmon JT, Tandon NN, Hoeg JM, Jamieson GA. Thrombin binding and response in platelets from patients with dyslipoproteinemias: increased stimulus-response coupling in type II hyperlipoproteinemia. Blood. 1986 Aug;68(2):498-505. PMID 3524709
- [Background] Wada H, Mori Y, Kaneko T, Wakita Y, Nakase T, Minamikawa K, Ohiwa M, Tamaki S, Tanigawa M, Kageyama S, et al. Elevated plasma levels of vascular endothelial cell markers in patients with hypercholesterolemia. Am J Hematol. 1993 Oct;44(2):112-6. doi: 10.1002/ajh.2830440208. PMID 8266915
- [Background] Davi G, Romano M, Mezzetti A, Procopio A, Iacobelli S, Antidormi T, Bucciarelli T, Alessandrini P, Cuccurullo F, Bittolo Bon G. Increased levels of soluble P-selectin in hypercholesterolemic patients. Circulation. 1998 Mar 17;97(10):953-7. doi: 10.1161/01.cir.97.10.953. PMID 9529262
- [Background] Garlichs CD, John S, Schmeisser A, Eskafi S, Stumpf C, Karl M, Goppelt-Struebe M, Schmieder R, Daniel WG. Upregulation of CD40 and CD40 ligand (CD154) in patients with moderate hypercholesterolemia. Circulation. 2001 Nov 13;104(20):2395-400. doi: 10.1161/hc4501.099312. PMID 11705814
- [Background] Puccetti L, Pasqui AL, Pastorelli M, Bova G, Cercignani M, Palazzuoli A, Angori P, Auteri A, Bruni F. Time-dependent effect of statins on platelet function in hypercholesterolaemia. Eur J Clin Invest. 2002 Dec;32(12):901-8. doi: 10.1046/j.1365-2362.2002.01086.x. PMID 12534449
- [Background] Violi F, Calvieri C, Ferro D, Pignatelli P. Statins as antithrombotic drugs. Circulation. 2013 Jan 15;127(2):251-7. doi: 10.1161/CIRCULATIONAHA.112.145334. No abstract available. PMID 23319813
- [Background] Ray KK, Cannon CP, McCabe CH, Cairns R, Tonkin AM, Sacks FM, Jackson G, Braunwald E; PROVE IT-TIMI 22 Investigators. Early and late benefits of high-dose atorvastatin in patients with acute coronary syndromes: results from the PROVE IT-TIMI 22 trial. J Am Coll Cardiol. 2005 Oct 18;46(8):1405-10. doi: 10.1016/j.jacc.2005.03.077. PMID 16226162
- [Background] Cipollone F, Mezzetti A, Porreca E, Di Febbo C, Nutini M, Fazia M, Falco A, Cuccurullo F, Davi G. Association between enhanced soluble CD40L and prothrombotic state in hypercholesterolemia: effects of statin therapy. Circulation. 2002 Jul 23;106(4):399-402. doi: 10.1161/01.cir.0000025419.95769.f0. PMID 12135935
- [Background] Undas A, Brummel-Ziedins KE, Potaczek DP, Stobierska-Dzierzek B, Bryniarski L, Szczeklik A, Mann KG. Atorvastatin and quinapril inhibit blood coagulation in patients with coronary artery disease following 28 days of therapy. J Thromb Haemost. 2006 Nov;4(11):2397-404. doi: 10.1111/j.1538-7836.2006.02165.x. Epub 2006 Aug 14. PMID 16907931
- [Background] Pawelczyk M, Chmielewski H, Kaczorowska B, Przybyla M, Baj Z. The influence of statin therapy on platelet activity markers in hyperlipidemic patients after ischemic stroke. Arch Med Sci. 2015 Mar 16;11(1):115-21. doi: 10.5114/aoms.2015.49216. Epub 2015 Mar 14. PMID 25861297
- [Background] Pignatelli P, Carnevale R, Pastori D, Cangemi R, Napoleone L, Bartimoccia S, Nocella C, Basili S, Violi F. Immediate antioxidant and antiplatelet effect of atorvastatin via inhibition of Nox2. Circulation. 2012 Jul 3;126(1):92-103. doi: 10.1161/CIRCULATIONAHA.112.095554. Epub 2012 May 21. PMID 22615342
- [Background] Blom DJ, Hala T, Bolognese M, Lillestol MJ, Toth PD, Burgess L, Ceska R, Roth E, Koren MJ, Ballantyne CM, Monsalvo ML, Tsirtsonis K, Kim JB, Scott R, Wasserman SM, Stein EA; DESCARTES Investigators. A 52-week placebo-controlled trial of evolocumab in hyperlipidemia. N Engl J Med. 2014 May 8;370(19):1809-19. doi: 10.1056/NEJMoa1316222. Epub 2014 Mar 29. PMID 24678979
- [Background] Sabatine MS, Giugliano RP, Wiviott SD, Raal FJ, Blom DJ, Robinson J, Ballantyne CM, Somaratne R, Legg J, Wasserman SM, Scott R, Koren MJ, Stein EA; Open-Label Study of Long-Term Evaluation against LDL Cholesterol (OSLER) Investigators. Efficacy and safety of evolocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1500-9. doi: 10.1056/NEJMoa1500858. Epub 2015 Mar 15. PMID 25773607
- [Background] Writing Committee; Lloyd-Jones DM, Morris PB, Ballantyne CM, Birtcher KK, Daly DD Jr, DePalma SM, Minissian MB, Orringer CE, Smith SC Jr. 2016 ACC Expert Consensus Decision Pathway on the Role of Non-Statin Therapies for LDL-Cholesterol Lowering in the Management of Atherosclerotic Cardiovascular Disease Risk: A Report of the American College of Cardiology Task Force on Clinical Expert Consensus Documents. J Am Coll Cardiol. 2016 Jul 5;68(1):92-125. doi: 10.1016/j.jacc.2016.03.519. Epub 2016 Apr 1. No abstract available. PMID 27046161
- [Background] Leoncini M, Toso A, Maioli M, Angiolillo DJ, Giusti B, Marcucci R, Abbate R, Bellandi F. High-dose atorvastatin on the pharmacodynamic effects of double-dose clopidogrel in patients undergoing percutaneous coronary interventions: The ACHIDO (Atorvastatin and Clopidogrel HIgh DOse in stable patients with residual high platelet activity) study. JACC Cardiovasc Interv. 2013 Feb;6(2):169-79. doi: 10.1016/j.jcin.2012.09.013. PMID 23428009
- [Background] Leoncini M, Toso A, Maioli M, Angiolillo DJ, Giusti B, Marcucci R, Abbate R, Bellandi F. Pharmacodynamic effects of adjunctive high dose atorvastatin on double dose clopidogrel in patients with high on-treatment platelet reactivity depending on diabetes mellitus status. J Thromb Thrombolysis. 2014 May;37(4):427-34. doi: 10.1007/s11239-013-0966-0. PMID 23852152
- [Background] Sikora J, Kostka B, Marczyk I, Krajewska U, Chalubinski M, Broncel M. Effect of statins on platelet function in patients with hyperlipidemia. Arch Med Sci. 2013 Aug 30;9(4):622-8. doi: 10.5114/aoms.2013.36905. Epub 2013 Aug 8. PMID 24049520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evolocumab | Placebo
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Due to Covid-19 pandemic, the trial was prematurely terminated | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients who have a clinical diagnosis of familial hypercholesterolemia and are referred for treatment with PCSK9 inhibitor, with LDL cholesterol levels ≥70 mg/dl on baseline treatment with statins and/or ezetimibe or intolerant to statin and/or ezetimibe.
Groups:
- Total: Total of all reporting groups
Arm/Group | Evolocumab | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Adenosine Di-phosphate (ADP) Induced, P2Y12 Dependent and Arachidonic Acid Induced Platelet Activation (P2Y12 Reaction Units (PRU))
Description: ADP- or arachidonic acid-stimulated platelet aggregation as assessed by the commercially-available VerifyNow P2Y12 (VerifyNow PRUTest) will be performed. Unit: PRU
Time Frame: Day 7, Day 14, Day 21, Day 28, Day 84
Population: Adult male and female subjects who have a clinical diagnosis of familial hypercholesterolemia and referred for treatment with PCSK9 inhibitor, with LDL cholesterol levels ≥70 mg/dl on baseline treatment with statins and/or ezetimibe or intolerant to statin and/or ezetimibe. Of the four participants reported in this study, one participant per arm had ADP assessed by PRU Test (evolocumab and placebo arms) and one participant per arm had ADP assessed by Aspirin assay (evolocumab and placebo arms).
Measure: Number; unit: PRU
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 1 | 1
PRU
  P2Y12 Test, Day 7 | 266 | 216
  P2Y12 Test, Day 14 | 268 | 226
  P2Y12 test, Day 21 | 268 | 233
  P2Y12 Test, Day 28 | 276 | 225
  P2Y12 Test, Day 84 | 256 | 267

2. Primary Outcome: Adenosine Di-phosphate (ADP) Induced, P2Y12 Dependent and Arachidonic Acid Induced Platelet Activation (Aspirin Reaction Unit (ARU))
Description: ADP- or arachidonic acid-stimulated platelet aggregation as assessed by the commercially-available VerifyNow Aspirin assay (Accriva Diagnostics) will be performed. Unit: Aspirin Reaction Unit (ARU)
Time Frame: Day 7, Day 14, Day 21, Day 28, Day 84
Population: as for outcome 1
Measure: Number; unit: ARU
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 1 | 1
ARU
  Aspirin Test, Day 7 | 521 | 432
  Aspirin Test Day 14 | 608 | 401
  Aspirin Test, Day 21 | 533 | 490
  Aspirin Test, Day 28 | 530 | 512
  Aspirin Test, Day 84 | 406 | 386

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Evolocumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT03331666/Prot_SAP_004.pdf